CLINICAL TRIAL: NCT04063163
Title: A Randomized, Double-Blind, Multicenter, Phase III Study to Compare Efficacy and Safety of HLX10 in Combination With Chemotherapy in Previously Untreated Patients With ES-SCLC
Brief Title: A Phase III Study to Investigate Efficacy and Safety of HLX10 + Chemotherapy in Patients With ES-SCLC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Henlius Biotech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HLX10-005-SCLC301
Record Dates: First submitted 2019-08-17; First posted 2019-08-21 (Actual); Results first posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Extensive Stage Small Cell Lung Cancer
Keywords: Extensive Stage; Small Cell Lung Cancer; Anti-PD-1 Monoclonal Antibody
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Carboplatin; Etoposide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A (Experimental): HLX 10+chemotherapy (Carboplatin-Etoposide)
  Interventions: Drug: HLX10; Drug: carboplatin and etoposide
- B (Placebo Comparator): Placebo+chemotherapy (Carboplatin-Etoposide)
  Interventions: Drug: carboplatin and etoposide; Drug: placebo

INTERVENTIONS:
Drug: HLX10 — HLX10 is an innovative monoclonal antibody targeting PD-1，developed by Shanghai Henlius Biotech, Inc.
  Arms: A
Drug: carboplatin and etoposide — chemotherapeutics
Drug: placebo — placebo
  Arms: B

SUMMARY:
This is a randomized, double-blind, multicenter, phase III clinical study to compare the clinical efficacy and safety of HLX10+ Chemotherapy vs placebo+Chemotherapy in Previously Untreated Patients with Extensive Stage Small Cell Lung Cancer.

Eligible subjects in this study will be randomized to Arm A or Arm B at 2:1 ratio as follows:

Arm A (HLX10 arm): HLX10 + chemotherapy (Carboplatin-Etoposide) ; Arm B (placebo arm): Placebo + chemotherapy (Carboplatin-Etoposide); The three stratification factors for randomization include: PD-L1 expression level (negative, positive, not available), Brain metastasis (yes versus no), Age (≥ 65 years versus < 65 years)

DETAILED DESCRIPTION:
After screening, subjects meeting the inclusion criteria and none of the exclusion criteria will be enrolled. Included subjects will be treated with HLX10 or placebo in combination with chemotherapy once every 3 weeks, until disease progression, death, intolerable toxicity, withdrawal of informed consent, or occurrence of other reasons specified in the protocol (whichever occurs first).

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically diagnosed with ES-SCLC (according to the Veterans Administration Lung Study Group staging system).
* No prior systemic therapy for ES-SCLC
* Major organs are functioning well
* Participant must keep contraception

Exclusion Criteria:

* Histologically or cytologically confirmed mixed SCLC.
* Known history of severe allergy to any monoclonal antibody.
* Known hypersensitivity to carboplatin or etoposide.
* Pregnant or breastfeeding females.
* Patients with a known history of psychotropic drug abuse or drug addiction.
* Patients who have other factors that could lead to the early termination of this study based on the investigator's judgment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 585 (Actual)
Dates: Start 2019-09-12 (Actual); Primary Completion 2024-05-07 (Actual); Study Completion 2024-05-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- Institute for Personalized Medicine, Tbilisi, Georgia
- Wojew. Wielospecjalistyczne Centrum Onkologii i Traumatologi, Lodz, Poland
- Arkhangelsk Clinical Oncology Dispensary, Arkhangelsk, Russia
- Medipol Mega Hospital, Istanbul, Turkey (Türkiye)
- Komunalnyi zaklad Miska bahato, Dnipropetrovsk, Ukraine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang K, Shen Y, Hu C, Xu F, Wang Q, Gao Y, Zhou L. Population Pharmacokinetics and Exposure-Response Analysis of Serplulimab in Small Cell Lung Cancer Patients. Clin Transl Sci. 2025 Sep;18(9):e70322. doi: 10.1111/cts.70322. PMID 40932107
- [Derived] Zhu Y, Liu K, Qin Q, Zhu H. Serplulimab plus chemotherapy as first-line treatment for extensive-stage small-cell lung cancer: A cost-effectiveness analysis. Front Immunol. 2023 Jan 4;13:1044678. doi: 10.3389/fimmu.2022.1044678. eCollection 2022. PMID 36685541
- [Derived] Cheng Y, Han L, Wu L, Chen J, Sun H, Wen G, Ji Y, Dvorkin M, Shi J, Pan Z, Shi J, Wang X, Bai Y, Melkadze T, Pan Y, Min X, Viguro M, Li X, Zhao Y, Yang J, Makharadze T, Arkania E, Kang W, Wang Q, Zhu J; ASTRUM-005 Study Group. Effect of First-Line Serplulimab vs Placebo Added to Chemotherapy on Survival in Patients With Extensive-Stage Small Cell Lung Cancer: The ASTRUM-005 Randomized Clinical Trial. JAMA. 2022 Sep 27;328(12):1223-1232. doi: 10.1001/jama.2022.16464. PMID 36166026
- See also: Effect of First-Line Serplulimab vs Placebo Added to Chemotherapy on Survival in Patients With Extensive-Stage Small Cell Lung Cancer — https://pmc.ncbi.nlm.nih.gov/articles/PMC9516323/

RESULTS

PARTICIPANT FLOW:
Groups:
- Group A: HLX 10+chemotherapy (Carboplatin-Etoposide)
  HLX10: HLX10 is an innovative monoclonal antibody targeting PD-1，developed by Shanghai Henlius Biotech, Inc.
  carboplatin and etoposide: chemotherapeutics
- Group B: Placebo+chemotherapy (Carboplatin-Etoposide)
  carboplatin and etoposide: chemotherapeutics
  placebo: placebo
Period: Overall Study
Arm/Group | Group A | Group B
Started | 389 | 196
Completed | 77 | 12
Not Completed | 312 | 184
Not completed — Death | 281 | 166
Not completed — Lost to Follow-up | 12 | 8
Not completed — Withdrawal by Subject | 19 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Total
Number analyzed (Participants) | 389 | 196 | 585
Age, Continuous [Mean (Full Range); unit: years] | 63 [28 to 76] | 62 [31 to 83] | 62 [28 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 72 | 164 | 236
  Male | 317 | 32 | 349
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 262 | 139 | 401
  Non-Asian | 127 | 57 | 184
Smoking history [Count of Participants; unit: Participants]
  Never smoker | 81 | 35 | 116
  Current smoker | 102 | 48 | 150
  Former smoker | 206 | 113 | 319

OUTCOME MEASURES:

1. Primary Outcome: OS
Description: Overall survival (OS)
Time Frame: The period from randomization through death regardless of causality (up to approximately 56 months)
Population: Analyses of the primary efficacy endpoint is based on the ITT. The ITT Population comprises all participants to whom study intervention has been randomized.
Measure: Median (95% Confidence Interval); unit: month
Groups:
- A Groups: HLX10+chemotherapy (Carboplatin-Etoposide)
- B Groups: Placebo+chemotherapy (Carboplatin-Etoposide)
Arm/Group | A Groups | B Groups
Number analyzed (Participants) | 389 | 196
month | 15.77 [13.897 to 17.413] | 11.10 [9.955 to 12.353]
Statistical Analysis 1: Comparison: A Groups vs B Groups; Defined as a period from randomization through death regardless of causality. Data of patients without a death record will be censored on the last known survival date. COX proportional risk model will be used to estimate HR and its 95% confidence interval (CI); the Kaplan-Meier method will be used to estimate the median, and the Kaplan-Meier curve will be plotted; Test type: Superiority; p < 0.001, Log Rank; Hazard Ratio (HR) = 0.62, 95% CI 2-sided [0.496 to 0.763]

2. Secondary Outcome: Progression Free Survival (PFS) Assessed by IRRC According to RECIST 1.1
Description: PFS is defined as a period from randomization initiation to the first documentation of PD or death regardless of causality (whichever occurs first).
Time Frame: From randomization initiation to the first documentation of PD or death regardless of causality, whichever occurs first (up to approximately 56 months).
Population: Analysis of PFS is based on ITT.
Measure: Median (95% Confidence Interval); unit: month
Arm/Group | A Groups | B Groups
Number analyzed (Participants) | 389 | 196
month | 5.82 [5.552 to 6.932] | 4.34 [4.205 to 4.435]
Statistical Analysis 1: Comparison: A Groups vs B Groups; Test type: Superiority; p = 0.001, Log Rank; Hazard Ratio (HR) = 0.47, 95% CI 2-sided [0.381 to 0.576]

3. Secondary Outcome: Objective Response Rate
Description: The ORR is defined as the proportion of subjects with a best overall response of CR or PR, according to RECIST 1.1. The best overall response will be defined as the best response across all time points in the order of CR, PR, SD, PD, and not NE.
Time Frame: From baseline until PR or CR, whichever occurs first (up to approximately 56 months)
Population: ORR is analyzed based on ITT.
Measure: Count of Participants; unit: Participants
Arm/Group | A Groups | B Groups
Number analyzed (Participants) | 389 | 196
Participants | 268 | 115

4. Secondary Outcome: Duration of Response
Description: DOR is defined as a period from the first documentation of response (CR or PR) through the first documentation of PD or death (whichever occurs first).
Time Frame: From the first documentation of response (CR or PR) through the first documentation of PD or death, whichever occurs first (up to approximately 56 months).
Population: DOR is analyzed based on ITT.
Measure: Median (95% Confidence Interval); unit: month
Arm/Group | A Groups | B Groups
Number analyzed (Participants) | 389 | 196
month | 6.80 [5.520 to 8.345] | 4.17 [3.055 to 4.205]

ADVERSE EVENTS:
Time Frame: From ICF until 90 days after the last study treatment (up to approximately 56 months).
Description: All AEs and treatment emergent AEs are recorded from the time of signing the ICF until 90 days after the last study treatment. If a subject starts a new antineoplastic therapy during the AE collection period, only information on AEs related to study treatment are collected after the new antineoplastic therapy.
Arm/Group | Group A | Group B
All-Cause Mortality (participants affected / at risk) | 224/389 | 140/196
Serious Adverse Events (participants affected / at risk) | 146/389 | 71/196
Other Adverse Events (participants affected / at risk) | 367/389 | 187/196
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group A (N=389) | Group B (N=196)
platelet count decreased (Blood and lymphatic system disorders) | 25 | 15
Neutrophil count decreased (Investigations) | 17 | 18
Neutrophil count decreased (Investigations) | 17 | 11
Alanine aminotransferase increased (Investigations) | 6 | 1
Aspartate aminotransferase increased (Investigations) | 3 | 0
Blood ketone body increased (Investigations) | 1 | 0
Fibrin D dimer increased (Investigations) | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0
Red blood cell count decreased (Investigations) | 1 | 0
Disease progression (General disorders) | 29 | 19
Death (Gastrointestinal disorders) | 11 | 7
Pyrexia (General disorders) | 4 | 2
Sudden death (General disorders) | 3 | 0
Asthenia (General disorders) | 0 | 3
Fatigue (General disorders) | 1 | 1
Non-cardiac chest pain (General disorders) | 1 | 1
Multiple organ dysfunction syndrome (General disorders) | 1 | 0
General physical health deterioration (General disorders) | 1 | 0
Pneumonia (Infections and infestations) | 14 | 7
COVID-19 (Infections and infestations) | 5 | 1
Septic shock (Infections and infestations) | 2 | 1
COVID-19 pneumonia (Infections and infestations) | 1 | 1
Device related infection (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 1 | 0
Lip infection (Infections and infestations) | 1 | 0
Lung abscess (Infections and infestations) | 1 | 0
Meningoencephalitis herpetic (Infections and infestations) | 1 | 0
Pneumonia bacterial (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Intracranial infection (Infections and infestations) | 0 | 1
Pneumonia aspiration (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Viral infection (Infections and infestations) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 11 | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 11 | 4
Leukopenia (Blood and lymphatic system disorders) | 9 | 3
Anaemia (Blood and lymphatic system disorders) | 6 | 5
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 3
Myelosuppression (Blood and lymphatic system disorders) | 1 | 0
Agranulocytosis (Blood and lymphatic system disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 4
Hyperglycaemia (Metabolism and nutrition disorders) | 5 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 2
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 2 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 3 | 0
Intestinal obstruction (Gastrointestinal disorders) | 2 | 1
Anal fissure (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Immune-mediated pancreatitis (Gastrointestinal disorders) | 1 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Immune-mediated encephalitis (Nervous system disorders) | 2 | 0
Cerebral infarction (Nervous system disorders) | 1 | 1
Aphasia (Nervous system disorders) | 1 | 0
Cognitive disorder (Nervous system disorders) | 1 | 0
Diabetic hyperosmolar coma (Nervous system disorders) | 1 | 0
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 1 | 0
Lacunar infarction (Nervous system disorders) | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0
Neurotoxicity (Nervous system disorders) | 1 | 0
Peripheral sensorimotor neuropathy (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 2 | 0
Angina pectoris (Cardiac disorders) | 1 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Cardiac failure acute (Cardiac disorders) | 1 | 0
Cardiopulmonary failure (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1
Cardiac tamponade (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Supraventricular extrasystoles (Cardiac disorders) | 0 | 1
Drug-induced liver injury (Hepatobiliary disorders) | 2 | 2
Hepatic function abnormal (Hepatobiliary disorders) | 2 | 0
Immune-mediated hepatitis (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 1
Hepatic lesion (Hepatobiliary disorders) | 0 | 1
Jaundice (Hepatobiliary disorders) | 0 | 1
Embolism (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
Venous thrombosis limb (Vascular disorders) | 1 | 0
Aortic arteriosclerosis (Vascular disorders) | 0 | 1
Aortic dissection rupture (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1
Embolism arterial (Vascular disorders) | 0 | 1
Hypovolaemic shock (Vascular disorders) | 0 | 1
Superior vena cava syndrome (Vascular disorders) | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0
Postoperative thrombosis (Injury, poisoning and procedural complications) | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Sternal fracture (Injury, poisoning and procedural complications) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 2 | 0
Ureterolithiasis (Renal and urinary disorders) | 1 | 0
Renal impairment (Renal and urinary disorders) | 0 | 1
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Anaphylactic reaction (Immune system disorders) | 1 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0
Vision blurred (Eye disorders) | 1 | 0
Panic disorder (Psychiatric disorders) | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group A (N=389) | Group B (N=196)
Anaemia (Blood and lymphatic system disorders) | 279 | 139
Neutropenia (Blood and lymphatic system disorders) | 115 | 59
Leukopenia (Blood and lymphatic system disorders) | 93 | 39
Thrombocytopenia (Blood and lymphatic system disorders) | 70 | 27
Neutrophil count decreased (Investigations) | 217 | 96
White blood cell count decreased (Investigations) | 205 | 98
Platelet count decreased (Investigations) | 157 | 85
Alanine aminotransferase increased (Investigations) | 71 | 37
Lymphocyte count decreased (Investigations) | 70 | 29
Aspartate aminotransferase increased (Investigations) | 62 | 33
Blood alkaline phosphatase increased (Investigations) | 48 | 17
Blood lactate dehydrogenase increased (Investigations) | 43 | 18
Weight decreased (Investigations) | 41 | 18
Weight increased (Investigations) | 43 | 14
Gamma-glutamyltransferase increased (Investigations) | 39 | 13
Blood cholesterol increased (Investigations) | 36 | 4
Blood bilirubin increased (Investigations) | 20 | 12
Blood creatinine increased (Investigations) | 20 | 10
Decreased appetite (Metabolism and nutrition disorders) | 109 | 56
Hyponatraemia (Metabolism and nutrition disorders) | 95 | 26
Hypoalbuminaemia (Metabolism and nutrition disorders) | 73 | 29
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 65 | 24
Hypokalaemia (Metabolism and nutrition disorders) | 58 | 14
Hyperglycaemia (Metabolism and nutrition disorders) | 50 | 15
Hypercholesterolaemia (Metabolism and nutrition disorders) | 44 | 19
Hyperuricaemia (Metabolism and nutrition disorders) | 41 | 17
Hypocalcaemia (Metabolism and nutrition disorders) | 40 | 10
Hypomagnesaemia (Metabolism and nutrition disorders) | 33 | 9
Hypochloraemia (Metabolism and nutrition disorders) | 29 | 11
Hypoproteinaemia (Metabolism and nutrition disorders) | 31 | 8
Hyperlipidaemia (Metabolism and nutrition disorders) | 23 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 20 | 5
Nausea (Gastrointestinal disorders) | 140 | 86
Constipation (Gastrointestinal disorders) | 94 | 58
Vomiting (Gastrointestinal disorders) | 78 | 58
Diarrhoea (Gastrointestinal disorders) | 38 | 13
Alopecia (Skin and subcutaneous tissue disorders) | 211 | 111
Rash (Skin and subcutaneous tissue disorders) | 30 | 8
Pyrexia (General disorders) | 60 | 24
Asthenia (General disorders) | 45 | 26
Fatigue (General disorders) | 34 | 13
Non-cardiac chest pain (General disorders) | 21 | 17
Malaise (General disorders) | 26 | 9
Chest discomfort (General disorders) | 13 | 10
Cough (Respiratory, thoracic and mediastinal disorders) | 47 | 23
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 28 | 27
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 18 | 18
Productive cough (Respiratory, thoracic and mediastinal disorders) | 19 | 10
Back pain (Musculoskeletal and connective tissue disorders) | 33 | 16
Arthralgia (Musculoskeletal and connective tissue disorders) | 33 | 13
Pain in extremity (Musculoskeletal and connective tissue disorders) | 31 | 14
Hypothyroidism (Endocrine disorders) | 64 | 7
Hyperthyroidism (Endocrine disorders) | 45 | 6
Urinary tract infection (Infections and infestations) | 25 | 13
Pneumonia (Infections and infestations) | 27 | 10
Dizziness (Nervous system disorders) | 28 | 10
Headache (Nervous system disorders) | 21 | 12
Insomnia (Psychiatric disorders) | 43 | 17
Proteinuria (Renal and urinary disorders) | 27 | 12
Sinus tachycardia (Cardiac disorders) | 21 | 6
Hypertension (Vascular disorders) | 16 | 11
Hepatic function abnormal (Hepatobiliary disorders) | 11 | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-30): https://cdn.clinicaltrials.gov/large-docs/63/NCT04063163/Prot_SAP_000.pdf